CLINICAL TRIAL: NCT05078762
Title: Immersive Virtual Reality in Simulation-based Bronchoscopy Training - a Randomized Trial
Brief Title: Immersive Virtual Reality in Simulation-based Bronchoscopy Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen Academy for Medical Education and Simulation (Other)
Responsible Party: Principal Investigator, Annarita Ghosh Andersen, Principal investigator, Copenhagen Academy for Medical Education and Simulation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: iVRBronch
Record Dates: First submitted 2021-09-22; First posted 2021-10-14 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Virtual Reality; Medical Education
Keywords: Bronchoscopy Training; Immersive Simulation Training

STUDY DESIGN:
Intervention Model Description: Randomization is performed online using SealedEnvelope™ (Sealed Envelope ltd, London, UK) before the start of the trial. The participants are stratified by sex (man/woman) as this has been seen to influence skills acquisition during the early part of in the learning curve
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants will not be blinded to the main investigator, as this is impossible due to the nature of the trial. The statistical analysis will be performed blinded and by someone other than the principal investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iVR (Experimental): The intervention group will train on a bronchoscopy simulator in an iVR environment with Virtual Reality Goggles (HTC IVE Pro Eye, HTC corporation, Taiwan) while using the bronchoscopy simulator.
  Interventions: Other: Immersive Virtual Reality
- Non iVR (No Intervention): The control group will train on a bronchoscopy simulator without VR goggles.

INTERVENTIONS:
Other: Immersive Virtual Reality — Training in an iVR environment with Virtual Reality Goggles while using the bronchoscopy simulator, while the control group will train without VR goggles.
  Other Names: iVR
  Arms: iVR

SUMMARY:
The purpose of this single-center randomized study is to investigate whether bronchoscopy training in an immersive Virtual Reality (iVR) environment will make the surgeon better at handling distractions and increase the quality of the bronchoscopy.

The participants will be stratified according to gender and randomized into two groups. Both groups will initially train on the bronchoscopy simulator without VR. Afterwards the intervention group will train in an iVR environment with Virtual Reality Goggles while using the bronchoscopy simulator, while the control group will train without VR goggles.

Afterwards both groups will be tested in the iVR environment in a test scenario

ELIGIBILITY:
Inclusion Criteria:

* Residents working in Denmark in thoracic surgery and pulmonary medicine
* Participants are required to have a medical license.

Exclusion Criteria:

* Previous participation in trials involving bronchoscopy training.
* Experience with independent bronchoscopy.
* No informed consent.
* Unable to speak Danish on a conversational level.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Based on a self-report form
Enrollment: 35 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Structured Progress | From beginning to end of each procedure, aprox. 30 minutes
  The systematic visualization and structured passage through the bronchial tree measured in points (0-18 points)
Procedure time | From beginning to end of each procedure, aprox. 30 minutes
  Time (seconds) from passing the vocal cords to retraction of the endoscope.

SECONDARY OUTCOMES:
Motor Bronchoscopy Skill Score | From beginning to end of each procedure, aprox. 30 minutes
  Objective and automatic composite score based on lower arm movement, measured with an Inertial Measurement Unit, and electromyography findings of hand and finger movement
Diagnostic completeness | From beginning to end of each procedure, aprox. 30 minutes
  The fraction in percent (%) of visited bronchial segments
Heart Rate Variability(LF/HF ratio) | From beginning to end of each procedure, aprox. 30 minutes
  The fraction between the low frequency and high frequency heart rate, measured as R-R intervals on an electrocardiogram for five minutes (17) Kubios HRV version 2.216 (Biosignal Analysis and Medical Group, Kuopio, Finland)
Eye movement measurements | From beginning to end of each procedure, aprox. 30 minutes
  Gaze direction (vector)
Eye movement measurements | From beginning to end of each procedure, aprox. 30 minutes
  Saccadic eye movements (gaze direction/time)
Eye movement measurements | From beginning to end of each procedure, aprox. 30 minutes
  Pupillary dilation (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Konge, Professor, MD, PHD, Study Chair — Copenhagen Academy for Medical Education and Simulation; Flemming Bjerrum, MD, PhD, Study Director — Copenhagen Academy for Medical Education and Simulation; Annarita G Andersen, BMed, Principal Investigator — Copenhagen Academy for Medical Education and Simulation
Locations (1):
- Copenhagen Academy for Medical Education and Simulation, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No